CLINICAL TRIAL: NCT04331392
Title: Remotely Delivered Environmental Enrichment Intervention for Traumatic Brain Injury: a Randomized Controlled Trial
Brief Title: Online Memory Intervention for Individuals with Traumatic Brain Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Ontario Neurotrauma Foundation (Other); Centre for Aging and Brain Health Innovation (Other)
Responsible Party: Principal Investigator, Robin Green, Principal Investigator, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-ABI-INFRA-1035
Record Dates: First submitted 2020-03-24; First posted 2020-04-02 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Brain Injuries, Traumatic; Brain Injury Traumatic Severe; Brain Injury Traumatic Moderate; Brain Injury, Chronic
Keywords: Environmental enrichment; spatial navigation; traumatic brain injury; neurorehabilitation; telerehabilitation; hippocampus
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injury, Chronic; Spatial Navigation

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the experimental intervention (allocentric navigation training) or the active control intervention (educational videos).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are blinded to whether they are completing the experimental or active control intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spatial navigation intervention (Experimental)
  Interventions: Behavioral: Spatial Navigation Intervention
- Educational Videos (Active Comparator)
  Interventions: Behavioral: Educational Videos

INTERVENTIONS:
Behavioral: Spatial Navigation Intervention — The 16-week intervention is completed daily, 5 days/week, remotely from home on a designated study website. Each week participants learn a new city through navigation tasks which increase in difficulty day-to-day and have a total of 4 levels of difficulty, with the goal of being able to independently navigate the city by the end of the week via Google Street View. Participants complete end-of-day multiple-choice tasks, testing what they learned with 3 types of allocentric questions: 1) predicting the next street/landmark, 2) distance judgement and 3) vector mapping. Participants also complete a map placement task, which involves reporting the locations of all studied landmarks/streets.
  Participants are presented with auditory rewards in the forms of short audio clips about landmarks, written encouragement in the form pop-ups (e.g., "Good work, keep it up!"), and coffee card rewards based on adherence to the intervention (e.g.,$5 bi-weekly if 100% of intervention is completed).
  Arms: Spatial navigation intervention
Behavioral: Educational Videos — The 16-week active control, remote video intervention is completed daily, 5 days a week by participants on a designated website. Participants placed in the active control group are trained on educational topics by watching videos of Ted Talks, to control for the effects of generalized environmental enrichment of the same dose as targeted navigation training. For each day of training, participants are asked to select between an option of 2 possible videos, watching a total of three videos per day. To ensure compliance and sufficient attention to the videos, at the end of each video, participants are asked to rate 5 aspects of the content (relevance, interest, comprehensibility, complexity, informative), and speaker (persuasiveness, quality of delivery, facial expression, convincingness, captivation), on a scale of 1 (lowest) to 5 (highest). Additionally, as with remote navigation participants, they are given written and monetary rewards.
  Arms: Educational Videos

SUMMARY:
This study will examine the behavioural and neurophysiological efficacy and feasibility of an online spatial navigation intervention for improving memory and brain health in individuals who have sustained moderate-severe traumatic brain injury.

DETAILED DESCRIPTION:
The memory impairments associated with moderate to severe traumatic brain injury can be debilitating to younger and older adults, and can prevent a person's return to work, school and social life. The "hippocampus" is a ubiquitously compromised memory brain structure in moderate-severe TBI. Unfortunately, not only does the hippocampus sustain the damage at the time of injury, but researchers have identified that it shows continued atrophy in the months and years following injury. The investigators has developed a promising behavioural intervention for arresting this shrinkage, enhancing the integrity of the hippocampus - and improving memory function. It entails engagement in novel, continuous and challenging allocentric spatial navigation, that is, learning new routes of cities, and making a map in one's head of those routes for 1 hour/day, 5 days per week for a period of 16 weeks. N=87 participants will be randomized to either the intervention group or an active control group that will watch 3 TedTalk videos per day, 5 days a week for the same duration. An MRI scan and cognitive measures focusing on memory and spatial navigation will be conducted before and after participation.

ELIGIBILITY:
Inclusion Criteria:

* acute care diagnosis of m-sTBI
* PTA of 24 hours or more and/or lowest GCS <13
* positive CT or MRI; (4) between 18 to 55 years of age
* fluency in English; (6) competency to provide informed consent or availability of a legal decision maker
* basic computer skills (use of internet/email, mouse and arrow keys)
* functional use of at least one upper extremity for computer use
* resident of Greater Toronto Area (to facilitate access to the MRI).

Exclusion Criteria:

* neurological disorder other than TBI (e.g., dementia, stroke)
* diagnosis of a neurodevelopmental disorder
* TBI sustained before age 18
* systemic comorbidities (e.g., lupus, diabetes)
* current diagnosis of aphasia
* presence of metal inside the body (e.g., surgical clips, pacemaker) leading to ineligibility for an MRI.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2018-10-30 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Imaging | Baseline and 1 week post-intervention.
  Efficacy of the intervention will be measured via Magnetic Resonance Imaging (MRI) to observe structural changes to the hippocampi and the integrity of associated white matter from baseline to 1 week post-intervention.
Change in Cognitive Map Formation Test (CMFT) (Medium transfer) performance, | Baseline and 1 week post-intervention.
  This assessment measures spatial memory and navigational ability through the formation and flexible use of a mental map of a new environment.
Change in Route Learning Navigation Test Battery - Different Approach Task (Medium transfer) performance. | Baseline and 1 week post-intervention.
  This task measures the ability to flexibly shift heading perspective.
Change in Path Integration Task (Medium transfer) performance. | Baseline and 1 week post-intervention.
  This task also assesses the ability to flexibly shift heading perspective, as well as path integration through a series of turns initiated by the participant walking through a maze.
Change in Memory Image Completion Task (MIC) (Far transfer) performance | Baseline and 1 week post-intervention.
  This task assesses the tendency for pattern completion processes of learned scenes.
Change in Mnemonic Similarity Test (MST) (Far transfer) performance | Baseline and 1 week post-intervention.
  This task reflects mnemonic discrimination ability that requires pattern separation by testing memory performance of images of everyday objects
Navigational abilities (near-transfer) | Measured throughout the completion of the 16-week spatial navigation intervention.
  To assess improvements to navigation-related, within-task intervention components, the following measures are collected for navigation training patients: 1) spatial learning ability based on end-of-day questions; 2) overall spatial ability improvement based on the difference in performance of end-of-week end-of-day questions, between earlier to later weeks of training; 3) independent navigation ability improvement Streetview-only reverse, alternate, and blocked routes, based on differences in performance between earlier to later weeks of training; and 4) cognitive map formation ability, based on differences in end-of-week performance between earlier and later weeks of training.
Change in Navigational Strategies Questionnaire score (medium transfer) | Baseline and 1 week post-intervention.
  Questionnaire measuring self-reported competence in cognitive mapping of routes and large-scale environments, and the formation of survey knowledge based on allocentric or environment-centered frames of reference. Questionnaire contains 14 questions with varying answers. Each response has an answer corresponding to a map-based navigation strategy or characteristic and one corresponding to a non-map/scene-based strategy. The mapping tendency is calculated as the difference between the number of map-based answers and non-map-based answers. Some questions have a third alternative, which is not coded. Final scores range from +14 to -14; the more positive, the more map-based navigation strategies a participant uses which is the better outcome.
Change in Santa Barbara Sense of Direction Scale score (medium transfer) | Baseline and 1-week post-intervention.
  Questionnaire measuring self-reported environmental spatial abilities. The responses are measured on a 7-point Likert scale (strongly agree = 1 - strongly disagree = 7), but is reversed for negative-worded questions. The final score is the average of all scores (between 1 and 7) where the higher the score, the better the perceived sense of direction. Increase in score is the better outcome.
Change in Everyday Memory Questionnaire score (far transfer) | Baseline and 1 week post-intervention.
  The test comprises statements regarding forgetting things and patients indicate how frequently the examples have occurred over the prior 3 months. The response options have the following scores: Once or less in the last month=0; More than once a month but less than once a week=1; About once a week=2; More that once a week or less than once a day=3; Once or more in a day=4.
  Final score for each participant is obtained by summing up all the scores from individual questions. Final score should range from 0-41, with higher the score, the better the memory. An increase in score is the better outcome.
Change in Digit Span score | Baseline and 1-week post-intervention.
  The test measures verbal working memory. Participants are asked to listen to a sequence of numbers and then to repeat the same sequence back to the examiner in order (forward span) or in reverse order (backward span). Each correct response is worth one point; with a maximum of 14 for each subscore series and for the total score, 28. The higher the score, the better verbal working memory. An increase in score is the better outcome.
Change in Visual Spatial Span score | Baseline and 1-week post-intervention.
  This task is a behavioral measure of visuospatial working memory capacity. In a sequence, the test administrator taps squares one at a time. The participant must then tap the squares in the same order that they were tapped by the administrator (for the forward variant) or in the reverse order (for backward variant). The number of boxes in the sequence increases from two at the start of the test, to nine at the end and the sequence. Each correct response is worth one point, up to a maximum of 44 points. The higher the score, the better memory. An increase in score is the better outcome.
Change in Sustained Attention to Response Test (SART) scores | Baseline and 1-week post-intervention.
  This is a Go/No-Go task measuring attention where participants view a computer monitor on which a random series of single digits are presented at the regular rate of 1 per 1.15 seconds. The task is to press a single response key following each presentation with the exception of a nominated No-Go digit, to which no response should be made. Performance is measured by calculating the number of errors of commission (inappropriately responding to a No-Go stimulus), errors of omission (inappropriately failing to respond to a Go stimulus) and reaction time to Go stimuli. Higher sustained attention should result in fewer errors of commission and omission, with shorter reaction time, which is the better outcome.
Change in Symbol Digit Modalities Test (SDMT) score | Baseline and 1-week post-intervention.
  The SDMT is a measure of information processing speed. This measure involves a coding key consisting of 9 abstract symbols, each paired with a number ranging from 1 to 9. The subject is required to scan the key and write down the number corresponding to each symbol as fast as possible. The score is the number of correctly coded items from 0-110 in 90 seconds, the higher the score the better the information processing speed. Higher score is the better outcome.
Change in the flanker inhibitory control and attention test score | Baseline and 1-week post-intervention.
  This test measures inhibitory control and selective attention. Participants are required to indicate the left-right orientation of a centrally presented stimulus while inhibiting attention to the potentially incongruent stimuli that surround it (i.e., the flankers, typically two on either side). A composite score of accuracy and reaction time is provided; the greater the score, the better attentional capacity. An increase in this score is the better outcome.
Change in the dimensional change card sort test score | Baseline and 1-week post-intervention.
  The test measures executive function. Participants sort a series of bivalent test cards, first according to one dimension (e.g., color), and then according to the other (e.g., shape), A composite score of accuracy and reaction time is provided; the greater the score, the better executive function performance reflecting high accuracy and short reaction time. Increase in score is the better outcome.
Change in pattern comparison processing speed test score | Baseline and 1-week post-intervention.
  The test measures information processing speed. Participants are asked to identify whether two visual patterns are the "same" or "not the same" by pressing respective button on the keyboard. Patterns were either identical or varied on one of three dimensions: color, adding/taking something away, or one versus many. Scores reflected the number of correct items (of a possible 130) completed in 90 seconds. The greater the score, the faster the processing speed. Increase in score is the better outcome.
Change in picture sequence memory test score | Baseline and 1-week post-intervention.
  The test measures episodic memory. Participant is presented with task stimuli: a sequence of pictured objects and activities related to a central theme (e.g. "working on the farm," "playing at the park,"). Participant must remember the specific order and reproduce it by placing the pictures in the correct temporal order. The score is derived from the cumulative number of adjacent pairs of pictures remembered correctly over the 3 trials. Higher score reflects better performance on task and thereby better episodic memory, which is the better outcome.
Change in Rey Auditory Verbal Learning Test (RAVLT) performance | Baseline and 1-week post-intervention.
  RAVLT measures verbal memory. Test administrator reads a list of 15 words at a rate of one per second. The patient's task is to repeat all the words he or she can remember, in any order. This procedure is carried out a total of five times. Then the examiner presents a second list of 15 words, allowing the patient only one attempt at recall. Immediately following this, the patient is asked to remember as many words as possible from the first list. A number of scores can be derived from the test including Immediate score (the sum of scores from 5 first trials), Learning score (the score of Trial 5 minus the score of Trial 1) and Forgetting score (the score of Trial 5 minus score of the delayed recall). The better outcomes would be increases in Immediate and Learning scores, decrease in Forgetting score.
Change in Rey Visual Design Learning Test (RVDLT) performance | Baseline and 1-week post-intervention.
  RVDLT measures memory for nonverbal material. Participants are asked to memorize 15 simple visual items that are presented one by one at a rate of 2 seconds per item. Then, they are asked to draw as many test items as can be remembered. This procedure is repeated four more times. After a 15-20 minutes delay, participants are asked again to draw as many items as possible. In the Recognition phase, a set of 30 visual items containing the test items shown before and 15 items not shown before are presented in random order, participants now have identify the ones shown before in the trials. A number of scores can be derived from the test including free recall score (the sum of scores from 5 first trials), Learning score (the score of Trial 5 minus the score of Trial 1) and Delayed Recall score (the score of Trial 6, after 15-20 minute delay). The better outcome would be an increase in these scores, reflecting an improvement in memory.

SECONDARY OUTCOMES:
Feasibility: Recruitment rate | Collected during recruitment
  Determined by dividing the number of patients consented by the number of eligible patients approached. Rate closer to 1 is desired.
Feasibility: Retention rate | Collected during recruitment and 1 week post-follow-up
  Determined by dividing the number of consented patients at baseline by the number of consented patients retained at follow-up. Factors influencing retention (e.g., medical status) will be reported as percentages. Rate closer to 1 is desired.
Feasibility: Compliance rate | Collected during each of the 80 session (5 sessions/week, 16 weeks)
  Determined by calculating the percentage of patients adhering to at least 80% of the training protocol. Compliance rates to be computed for individual participants weekly, and for full cohort at end of study. Rate closer to 100% is desired.
  Factors influencing recruitment, retention and completion will be documented and reported as percentages.
Feasibility: semi-structured interview | 1 week post-intervention
  A semi-structured interview will be administered at post-intervention assessment to ascertain experience with the intervention, and any barriers and facilitation to participation. A qualitative thematic analysis will be applied and key themes will be reported on.
Change in How Much Is Too Much scale score | At the end of each of the 16 weeks
  This scale was developed by our group to quantify a patient's experience of cognitive, somatic and emotional burden in response to completing a cognitive intervention. A list of 26 symptoms will be provided, and the patient will be asked to select whether they have experienced each symptom "Less than before my session today" (=-1); "The same as before my session today" (=0); "I did not have this symptom at all today" (=0); "More than before my session today (=1); "Much more than before my session today" (=2).
  By scoring each response according to the number in brackets, and averaging the numbers for all patients per symptom per week, we will evaluate whether participants experienced any particular symptom more often as a result of the intervention across the 16 weeks. Decrease in scores or maintaining a score of 0 week-to-week are the desired outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Robin E Green, PhD; CPsych, Principal Investigator — Toronto Rehabilitation Institute; Asaf Gilboa, PhD, Principal Investigator — Baycrest Health Sciences
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data will be shared that underlie the results reported in the first empirical article published on this study article, after deidentification (text, tables, figures, and appendices). Due to sensitivity of patient information and to reduce risk of identification, demographic information will be limited to age band, gender and highest education level achieved.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data pertaining to primary outcomes will become available within one year of publication of the first empirical paper. It would be available until September 2028.
Access Criteria: Data will be made openly and publicly available on Dryad Digital Repository. Upon reasonable request, further data can be made available to researchers who provide a methodologically sound proposal for any analyses (e.g. meta-analysis) that work to achieve aims in the approved proposal. Proposals should be directed to robin.green@uhn.ca or agilboa@research.baycrest.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Corrow JC, Corrow SL, Lee E, Pancaroglu R, Burles F, Duchaine B, Iaria G, Barton JJS. Getting lost: Topographic skills in acquired and developmental prosopagnosia. Cortex. 2016 Mar;76:89-103. doi: 10.1016/j.cortex.2016.01.003. Epub 2016 Jan 22. PMID 26874939
- [Background] Wiener JM, Carroll D, Moeller S, Bibi I, Ivanova D, Allen P, Wolbers T. A novel virtual-reality-based route-learning test suite: Assessing the effects of cognitive aging on navigation. Behav Res Methods. 2020 Apr;52(2):630-640. doi: 10.3758/s13428-019-01264-8. PMID 31236900
- [Background] Persson J, Herlitz A, Engman J, Morell A, Sjolie D, Wikstrom J, Soderlund H. Remembering our origin: gender differences in spatial memory are reflected in gender differences in hippocampal lateralization. Behav Brain Res. 2013 Nov 1;256:219-28. doi: 10.1016/j.bbr.2013.07.050. Epub 2013 Aug 9. PMID 23938766
- [Background] Vieweg P, Riemer M, Berron D, Wolbers T. Memory Image Completion: Establishing a task to behaviorally assess pattern completion in humans. Hippocampus. 2019 Apr;29(4):340-351. doi: 10.1002/hipo.23030. Epub 2018 Nov 23. PMID 30246900
- [Background] Vieweg P, Stangl M, Howard LR, Wolbers T. Changes in pattern completion--a key mechanism to explain age-related recognition memory deficits? Cortex. 2015 Mar;64:343-51. doi: 10.1016/j.cortex.2014.12.007. Epub 2014 Dec 29. PMID 25597525
- [Background] Stark SM, Yassa MA, Lacy JW, Stark CE. A task to assess behavioral pattern separation (BPS) in humans: Data from healthy aging and mild cognitive impairment. Neuropsychologia. 2013 Oct;51(12):2442-9. doi: 10.1016/j.neuropsychologia.2012.12.014. Epub 2013 Jan 9. PMID 23313292
- [Background] Sunderland, A., Harris, J. E., & Baddeley, A. D. (1983). Do laboratory tests predict everyday memory? A neuropsychological study. Journal of verbal learning and verbal behavior, 22(3), 341-357.
- [Background] Wiener, J., & Wolbers, T. (2018). Route Learning & Navigation Test Battery. Retrieved from osf.io/mx52y
- [Background] Brunec IK, Bellana B, Ozubko JD, Man V, Robin J, Liu ZX, Grady C, Rosenbaum RS, Winocur G, Barense MD, Moscovitch M. Multiple Scales of Representation along the Hippocampal Anteroposterior Axis in Humans. Curr Biol. 2018 Jul 9;28(13):2129-2135.e6. doi: 10.1016/j.cub.2018.05.016. Epub 2018 Jun 21. PMID 29937352
- [Background] Hegarty, M., Richardson, A. E., Montello, D. R., Lovelace, K., & Subbiah, I. (2002). Development of a self-report measure of environmental spatial ability. Intelligence, 30(5), 425-448
- [Derived] Belchev Z, Boulos ME, Rybkina J, Johns K, Jeffay E, Colella B, Ozubko J, Bray MJC, Di Genova N, Levi A, Changoor A, Worthington T, Gilboa A, Green R. Remotely delivered environmental enrichment intervention for traumatic brain injury: Study protocol for a randomised controlled trial. BMJ Open. 2021 Feb 11;11(2):e039767. doi: 10.1136/bmjopen-2020-039767. PMID 33574141